CLINICAL TRIAL: NCT00638625
Title: Pilot Study of Radiologic-Pathologic Correlation in Lung Tumors Based on Core Needle Biopsy
Brief Title: Correlation of X-ray and Pathology With Needle Biopsy of Lung Tumors
Status: Withdrawn | Type: Observational
Why Stopped: Due to specimen collection difficulties; this study has been terminated
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Ernest Scalzetti, MD, State University of New York - Upstate Medical University
Other Study IDs: SUNYUMU 5376
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Lung Neoplasm
Keywords: Needle biopsy; CT Scan; Lung Tumor; Lung Mass
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare the features that the pathologist sees, when examining a lung tumor under the microscope, to the way that the tumor appears on the computed tomography (CT) scan. Features of the tumor may include abnormal blood vessels and areas in which tumor cells are dying. The samples that are taken during the needle biopsy contain information from one small part of the tumor. The investigators believe that they can show where in the tumor the samples came from, based on the CT scans during the biopsy procedure. If the investigators can accurately determine where in the tumor their samples came from, they can compare the features of that part of the tumor, as seen on the CT images, to the features of that part of the tumor as seen under the microscope. This research study also will give the investigators an idea of how much the biopsy samples are distorted in the process of preparing them for examination under the microscope.

DETAILED DESCRIPTION:
Newer cross-sectional imaging methods allow improved visualization of anatomic detail-for example, high-resolution CT has a spatial resolution of less than 1 mm in all 3 dimensions. These imaging methods also provide a limited amount of physiologic information-for example, tumor perfusion as demonstrated by enhancement with intravenous contrast agents. Radiologic-pathologic correlation in the current era gives us the opportunity to work on a finer spatial scale and to take advantage of the additional physiologic information. Pathologic assessment of tissue has evolved at the same time. Tissue can be stained in the traditional way for microscopic evaluation but newer tools such as immunohistochemistry and, most recently, methods of molecular biology can be applied as well.

We are interested in radiologic-pathologic correlation in lung tumors. Tumors are known to be heterogeneous; we want to develop an approach that will allow us to explore their spatial organization. We cannot rely on surgical resection to provide tissue for pathologic evaluation, because the majority of lung lesions never come to resection. For example, only ~15% of lung cancer patients are surgical candidates. The remainder would be lost to the classical approach that depends on surgery. Percutaneous needle biopsy provides an alternative means of tissue sampling. This is a safe, effective and commonly used way to obtain samples of tissue ("core samples") from any given lung mass. The pathologist can process these core samples in the same way as a surgical specimen.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have a lung tumor that is likely to be malignant
* Subjects who have been referred for percutaneous needle biopsy
* The target lesion must be at least 10 mm in short-axis dimension.
* Subjects must have intravenous access.
* No history of significant allergy to intravenous contrast.
* Subjects must have sufficient renal function to receive intravenous contrast for enhancement of the CT images.

Exclusion Criteria:

* Vulnerable populations will be excluded.
* Subjects who lack the capacity to provide consent
* Subjects who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study subjects will be recruited among patients who are referred for percutaneous needle biopsy of a suspected malignant lesion in the lung. Consecutive patients who meet the eligibility criteria will be offered enrollment until the study accrual target has been met.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Determination of the accuracy of registration of contrast-enhanced CT images to the CT images that show the location of the core tissue sample

SECONDARY OUTCOMES:
Determination of the dimensional stability of the core tissue sample: whether, and if so, how much, the length of the core sample changes as it is processed

CONTACTS AND LOCATIONS:
Overall Officials: Ernest Scalzetti, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States